CLINICAL TRIAL: NCT05427747
Title: Meropenem vs Cefotaxime as Empirical Treatment of Spontaneous Bacterial Peritonitis :Prospective Randomized Clinical Trial
Brief Title: Meropenem vs Cefotaxime as Empirical Treatment of SBP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Taha Hussein Kawashty Abdelrahman, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Meropenem vs cefotaxime in SBP
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Cefotaxime; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cefotaxime (Experimental): ceotaxime 2g iv /8hr
  Interventions: Drug: cefotaxime
- meropenem (Experimental): meropenem 1g iv /8hr
  Interventions: Drug: cefotaxime

INTERVENTIONS:
Drug: cefotaxime — One group will be given cefotaxime and another group meropenem.
  The efficacy of antibiotic therapy will be checked with:
  * Follow-up paracentesis after 48 hours of initiation of empiric antibiotic treatment showing reduction in neutrophil count of at least 25% .
  * Decrease of peritoneal fluid PMN count to < 250 cells/μ at end of treatment and negative previously positive ascitic fluid culture.
  Other Names: meropenem

SUMMARY:
We aimed to evaluate whether meropenem is superior to cefotaxime for treatment of SBP empirically.

DETAILED DESCRIPTION:
Ascites is the most frequent complication of cirrhosis and represents a significant change for the patient because the impact on mortality and quality of life is important.

Spontaneous bacterial peritonitis (SBP) is a dreaded complication in patients with decompensated cirrhosis.

Spontaneous bacterial peritonitis (SBP) is the most frequent and life-threatening infection in patients with liver cirrhosis requiring prompt recognition and treatment. It is defined by the presence of >250 polymorphonuclear cells (PMN)/mm3 in ascites in the absence of an intra-abdominal source of infection or malignancy.

Spontaneous bacterial peritonitis carries a mortality rate of 30 to 70% in patients with end-stage liver and kidney disease.

Choice of antibiotic is dependent on type of microbes responsible for infection. Gram negative enteric bacteria are considered the most common pathogens responsible for SBP. This is the reason, 3rd generation cephalosporins are the recommended drugs of choice for treating SBP empirically. But recent studies have shown that Cephalosporins are effective only in 70% of community acquired and 56% of hospital acquired SBP.It is most likely due to changing bacterial pathogens of SBP over last two decades as now gram positive bacteria and multi drug resistance organism (MDRO) are increasingly being isolated in SBP. It is the consequence of undue, over the counter misuse of cephalosporins in community and frequent exposure of cirrhosis patients to these drugs during recurrent hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis patients with ascites Ascitic fluid PMN cell count >250/mm3 Age: 18:80

Exclusion Criteria:

* : history of abdominal surgery within 4 weeks, secondary peritonitis, tuberculous peritonitis, Malignant tumor, patients who use hormones or immunosuppressants, AIDS patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Response to treatment within 5 days | 5 days
  The response to therapy is defined as the reduction of polymorphonuclear leukocytes (PMN) count in ascitic fluid more than 25 % from baseline after 48 hours and as a PMN count in ascitic fluid less then 250/mm³ after 5 days

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Finci L, Mouraux S, Knuchel J, Bochatay L. [Initial management of new onset ascites in patient with cirrhosis]. Rev Med Suisse. 2017 Sep 6;13(573):1509-1515. French. PMID 28876707
- [Result] Sarwar S, Tarique S, Waris U, Khan AA. Cephalosporin resistance in community acquired spontaneous bacterial peritonitis. Pak J Med Sci. 2019 Jan-Feb;35(1):4-9. doi: 10.12669/pjms.35.1.17. PMID 30881387
- [Result] Wiest R, Krag A, Gerbes A. Spontaneous bacterial peritonitis: recent guidelines and beyond. Gut. 2012 Feb;61(2):297-310. doi: 10.1136/gutjnl-2011-300779. Epub 2011 Dec 6. No abstract available. PMID 22147550
- [Result] Ameer MA, Foris LA, Mandiga P, Haseeb M. Spontaneous Bacterial Peritonitis(Archived). 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448208/ PMID 28846337